CLINICAL TRIAL: NCT07336147
Title: Dostarlimab, Cisplatin and Etoposide in Combination With Radiotherapy in Sandwich Sequence for Small Cell Neuroendocrine Cervical Carcinoma (DICER Trial): Taiwanese Gynecologic Oncology Group (TGOG) 1012
Brief Title: Dostarlimab, Cisplatin and Etoposide in Combination With Radiotherapy in Sandwich Sequence for Small Cell Neuroendocrine Cervical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, LAI, CHYONG-HUEY, Taiwanese Gynecologic Oncology Group, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202501489A0
Record Dates: First submitted 2025-12-29; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Female
Keywords: dostarlimab; cisplatin; etoposide; cervical carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dostarlimab (Experimental): The planned dose of dostarlimab for this study is 500 mg every 3 weeks (Q3W) during chemoimmunotherapy phase. Based on the totality of data generated in the dostarlimab development program, either 500 mg Q3W or 1000 mg Q6W is the appropriate dose of dostarlimab for adults across all indications and regardless of tumor type.
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — The planned dose of dostarlimab for this study is 500 mg every 3 weeks (Q3W) during chemoimmunotherapy phase. Based on the totality of data generated in the dostarlimab development program, either 500 mg Q3W or 1000 mg Q6W is the appropriate dose of dostarlimab for adults across all indications and regardless of tumor type.

SUMMARY:
Add-on dostarlimab to chemoradiation with etoposide and cisplatin and radiotherapy can improve progression-free survival (PFS) compared with historical controls who were treated with chemoradiation alone in SCNECC

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are 20-70 years of age on the day of signing informed consent with histologically confirmed diagnosis of Previously untreated SCNECC IB2-IV or IB1 with LVSI or IVB with oligometastasis (only in one distant organ not more than 2 nodules which can be encompassed by RT) will be enrolled in this study.

   *A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to participate this trial should be informed that after the protocol treatment the ovarian function and child-bearing potential will be permanently lost and she has to follow the contraceptive guidance in Appendix 3 after enrollment through neoadjuvant chemoimmuntherapy period till external beam radiotherapy (EBRT) commences.
2. Have provided archival tumor tissue sample or newly obtained biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archival tissue. At least 5 punch biopsiesdof 3mm in diameter.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy for SCNECC including investigational agents prior to enrollment.
4. Has received prior pelvic radiotherapy.
5. Has received radical surgery for cervical cancer.
6. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
10. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
11. Has severe hypersensitivity (≥Grade 3) to dostarlimab and/or any of its excipients.
12. Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
13. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
14. Has an active infection requiring systemic therapy.
15. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
16. Has a known history of untreated Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection (for those with anti-HCV+, patients who ever HCV RNA positive should undergo 8-12 weeks direct acting agents (DAA) treatment and confirmed with HCV cure, defined as HCV RNA negative at week 12 post end-of-treatment). Note: Testing for Hepatitis B and Hepatitis C is required but the patient is eligible if well controlled.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Allergy: Participant cannot have history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies or fusion proteins, sensitivity to any of the study treatments or components thereof, or a history of drug or other allergy that contraindicates their participation.
19. Has had an allogenic tissue/solid organ transplant.
20. Participant has received a live vaccine within 30 days of planned start of study therapy. COVID-19 vaccines that do not contain live viruses are allowed. Note: mRNA and adenoviral-based COVID-19 vaccines are considered non-live.
21. Participant has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.

Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.

-

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-12-22 (Estimated); Study Completion 2030-12-22 (Estimated)

PRIMARY OUTCOMES:
Dostarlimab, with radiotherapy in sandwich sequence for small cell neuroendocrine cervical carcinoma. PFS at 2 years (from 57% to 75%) PFS is defined the date of starting chemotherapy with dostarlimab to the date of progression defined with RECIST 1.1 | 588 DAYS
  Add-on dostarlimab to chemoradiation with etoposide and cisplatin can prolong OS with acceptable tolerability and maintaining quality of life (QOL).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taiwan, Taiwan